CLINICAL TRIAL: NCT04732195
Title: A Pilot Study to Compare the Efficacy of Pilocarpine Microneedles With Iontophoresis Method for Sweat Induction in Healthy Human Subjects
Brief Title: Pilocarpine Microneedles for Sweat Induction (PMN-SI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Georgia Institute of Technology (Other)
Responsible Party: Principal Investigator, Lokesh Guglani, Associate Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00115911
Record Dates: First submitted 2021-01-25; First posted 2021-02-01 (Actual); Results first posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-04

CONDITIONS: Cystic Fibrosis
Keywords: Sweat test; Microneedle; Pilocarpine; Cystic fibrosis; Iontophoresis; Drug Delivery
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Pilocarpine microneedle patch (Experimental): Participants will receive in their left forearm the microneedle patch. Upon application to skin, the MNs penetrate into the skin's upper layers and dissolve in the interstitial fluid to release the loaded drugs. MN patches are painless and can be administered with little or no training.
  Interventions: Device: Pilocarpine microneedle patch
- Pilocarpine Iontophoresis (Active Comparator): Participants will receive in their right forearm the pilocarpine iontophoresis. Uses a gel disc containing Pilocarpine that drives the medication into the skin with a small electric current (iontophoresis) followed a 30-minute period of sweat collection.
  Interventions: Device: Pilocarpine Iontophoresis

INTERVENTIONS:
Device: Pilocarpine microneedle patch — Each microneedle (MN) patch contains an array of solid, water-soluble, micron-scale needles that encapsulate the medication (Pilocarpine). The patch form can be placed directly on the skin.
  Other Names: Microneedle patch
  Arms: Pilocarpine microneedle patch
Device: Pilocarpine Iontophoresis — Pilocarpine Iontophoresis is a process of transdermal pilocarpine delivery by use of a voltage gradient on the skin. An agar gel disc containing pilocarpine is placed under the electrodes which are connected to the Macroduct 3700 Sweat Inducer device.
  Arms: Pilocarpine Iontophoresis

SUMMARY:
The investigators want to test in this non-randomized clinical trial a new method of administrating Pilocarpine medicine into the skin during the Sweat testing process that does not use any electrical current.

DETAILED DESCRIPTION:
Sweat collection tests are done when a patient is suspected of having cystic fibrosis. This procedure for collection of sweat samples is called the Sweat Test and the measurement of sweat chloride concentration from the collected sweat sample is the gold standard for the diagnosis of Cystic Fibrosis.

When the sweat test is performed for patients in a hospital lab, the standard method uses a small electrical current to push pilocarpine medicine into the skin of the forearm, after which sweat is collected for testing. However, many people do not make enough sweat during this standard method of testing and have to come back for repeated testing. The investigators want to test a new method of putting Pilocarpine medicine into the skin during the Sweat testing process that does not use any electrical current.

The testing will be done once for every participant and no further follow up or additional testing is needed. The study team plans to invite healthy adults who are not taking any medicines to participate through a flyer posted in Emory Children's Center bulletin board. For those interested in participating, the study will be explained to them in detail and an informed consent will be obtained. The subjects will be asked to sit for 45 minutes on a chair as the study related procedures are completed on their arms. The right forearm will be used for pilocarpine iontophoresis method and the left forearm will be used for microneedle-based stimulation method for a period of 5 minutes. An additional microneedle control patch (without any Pilocarpine) will be placed on the left forearm to make sure that there are no skin changes from the microneedles. After the first 5 minutes, the sweat collection devices (Macroduct) will be placed on both forearms to collect sweat samples from each site. After the completion of this 30-minute collection phase, the Macroduct collectors will be removed by the study team and the subject testing will be complete. The study team will store the sweat samples to measure their chloride concentration at the end of the enrollment phase of the study.

This study will be conducted in a research room at Emory Children's Center and no compensation will be provided to the participants. At the end of the study, the research team will compare the two methods based on how much sweat was produced in each individual's arms with either of these methods. The results of this study will help to improve the current technique of sweat testing and help reduce the need for repeated testing in patients being evaluated for Cystic Fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Signed a written informed consent
* Not taking any medications
* No known medical diagnoses or chronic conditions

Exclusion Criteria:

* Age <18 years
* Family history of Cystic Fibrosis
* History of skin disorders (eczema, psoriasis etc.) that could prevent sweat testing on forearms
* Current medication use

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2022-03-17 (Actual); Study Completion 2022-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lokesh Guglani, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta - Egleston Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen JY, Li S, Silva GL, Chandler JD, Prausnitz MR, Guglani L. Sweat induction using Pilocarpine microneedle patches for sweat testing in healthy adults. J Cyst Fibros. 2024 Jan;23(1):112-119. doi: 10.1016/j.jcf.2023.04.014. Epub 2023 May 25. PMID 37236899

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 50 subjects provided informed consent for participation in this study. Participants had 2 different types of sweat collection method, one in each arm: the standard of care pilocarpine iontophoresis method on the left forearm and the pilocarpine microneedle patch method on the right forearm. The 50 subjects were able to undergo sweat testing on both forearms during their study visit.
Units Other Than Participants: sweat samples
Groups:
- Pilocarpine Microneedle Patch Method: Participants received in their left forearm the microneedle patch. Upon application to skin, the MNs penetrate into the skin's upper layers and dissolve in the interstitial fluid to release the loaded drugs. MN patches are painless and can be administered with little or no training.
  Pilocarpine microneedle patch: Each microneedle (MN) patch contains an array of solid, water-soluble, micron-scale needles that encapsulate the medication (Pilocarpine). The patch form can be placed directly on the skin.
- Pilocarpine Iontophoresis Method: Participants received in their right forearm the pilocarpine iontophoresis. Uses a gel disc containing Pilocarpine that drives the medication into the skin with a small electric current (iontophoresis) followed a 30-minute period of sweat collection.
  Pilocarpine Iontophoresis: Pilocarpine Iontophoresis is a process of transdermal pilocarpine delivery by use of a voltage gradient on the skin. An agar gel disc containing pilocarpine is placed under the electrodes which are connected to the Macroduct 3700 Sweat Inducer device.
Period: Overall Study
Arm/Group | Pilocarpine Microneedle Patch Method | Pilocarpine Iontophoresis Method
Started | 50; 50 sweat samples | 50; 50 sweat samples
Completed | 50; 50 sweat samples | 50; 50 sweat samples
Not Completed | 0; 0 sweat samples | 0; 0 sweat samples

BASELINE CHARACTERISTICS:
Population: A total of 50 subjects provided informed consent for participation in this study. Participants had 2 different types of sweat collection method, one in each arm: the standard of care pilocarpine iontophoresis method on the left forearm and the pilocarpine microneedle patch method on the right forearm. The 50 subjects were able to undergo sweat testing on both forearms during their study visit.
Units Other Than Participants: sweat samples
Groups:
- Total: Total of all reporting groups
Arm/Group | Pilocarpine Microneedle Patch Method | Pilocarpine Iontophoresis Method | Total
Number analyzed (Participants) | 50 | 50 | 50
Number analyzed (sweat samples) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (9.84) | 35 (9.84) | 35 (9.84)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: A total of 50 subjects provided informed consent for participation in this study. Participants had 2 different types of sweat collection method, one in each arm: the standard of care pilocarpine iontophoresis method on the left forearm and the pilocarpine microneedle patch method on the right forearm. The 50 subjects were able to undergo sweat testing on both forearms during their study visit.
  Participants
    Female | 34 | 34 | 68
    Male | 16 | 16 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: A total of 50 subjects provided informed consent for participation in this study. Participants had 2 different types of sweat collection method, one in each arm: the standard of care pilocarpine iontophoresis method on the left forearm and the pilocarpine microneedle patch method on the right forearm. The 50 subjects were able to undergo sweat testing on both forearms during their study visit.
  Participants
    Hispanic or Latino | 9 | 9 | 18
    Not Hispanic or Latino | 41 | 41 | 82
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 12 | 12 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 7 | 14
  White | 22 | 22 | 44
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 9 | 18
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 50
Sweat collection volume type [Number; unit: sweat samples]
  Adequate sweat collection (>15uL) | 44 | 43 | 87
  Insufficient sweat collection (<15uL) | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Amount of Sweat Collected
Description: Sweat weight in mg collected after application of Pilocarpine Microneedle patch was compared to the forearm of healthy adult subjects with that of standard of care method using pilocarpine iontophoresis
Time Frame: 45 min Post-intervention
Population: For purposes of this analysis only sweat samples with adequate volume were included from each of the participants.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Pilocarpine Microneedle Patch Method | Pilocarpine Iontophoresis Method
Number analyzed (Participants) | 44 | 43
mg | 41.2 (25.0) | 43.8 (32.3)

2. Secondary Outcome: Sweat Chloride Concentration
Description: Sweat chloride concentrations will be measured from the sweat samples obtained from the application of Pilocarpine Microneedle patch to the forearm of healthy adult subjects and compare them with measurements from standard of care method using pilocarpine iontophoresis.
Time Frame: 45 min Post-intervention
Population: For purposes of this analysis only sweat samples with adequate volume were included from each of the participants.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Pilocarpine Microneedle Patch Method | Pilocarpine Iontophoresis Method
Number analyzed (Participants) | 44 | 43
mmol/L | 31.2 (13.4) | 24.0 (13.2)

ADVERSE EVENTS:
Time Frame: All enrolled subjects were observed for a total period of 1 hour from the time consent was given and all testing and follow up evaluation completed.
Groups:
- Pilocarpine Microneedle Patch Method: Participants will receive in their left forearm the microneedle patch. Upon application to skin, the MNs penetrate into the skin's upper layers and dissolve in the interstitial fluid to release the loaded drugs. MN patches are painless and can be administered with little or no training.
  Pilocarpine microneedle patch: Each microneedle (MN) patch contains an array of solid, water-soluble, micron-scale needles that encapsulate the medication (Pilocarpine). The patch form can be placed directly on the skin.
- Pilocarpine Iontophoresis Method: Participants will receive in their right forearm the pilocarpine iontophoresis. Uses a gel disc containing Pilocarpine that drives the medication into the skin with a small electric current (iontophoresis) followed a 30-minute period of sweat collection.
  Pilocarpine Iontophoresis: Pilocarpine Iontophoresis is a process of transdermal pilocarpine delivery by use of a voltage gradient on the skin. An agar gel disc containing pilocarpine is placed under the electrodes which are connected to the Macroduct 3700 Sweat Inducer device.
Arm/Group | Pilocarpine Microneedle Patch Method | Pilocarpine Iontophoresis Method
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/95/NCT04732195/Prot_SAP_000.pdf